CLINICAL TRIAL: NCT04902183
Title: A Phase II Randomized, Single-blind Dose Study to Evaluate the Safety and Efficacy of Exosomes Overexpressing CD24 in 10^9 Dose Versus 10^10 Dose, for the Prevention of Clinical Deterioration in Patients With Moderate or Severe COVID-19
Brief Title: Safety and Efficacy of Exosomes Overexpressing CD24 in Two Doses for Patients With Moderate or Severe COVID-19
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Athens Medical Society (Other)
Collaborators: OBCTCD24 Ltd (Unknown); Elpen Pharmaceutical Co. Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NS3
Record Dates: First submitted 2021-05-21; First posted 2021-05-26 (Actual); Last update posted 2021-06-15 (Actual); Status verified 2021-06

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: This is a two arms study; one arm will receive 10^9 dose and the second arm will receive 10^10 dose of exosomes overexpressing CD24
Who Masked: Participant
Masking Description: The administrated dose will be unknown to the patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 10^9 dose of exosomes overexpressing CD24 (Experimental): The patients will receive the dose of 10^9 exosomes overexpressing CD24
  Interventions: Drug: CovenD24
- 10^10 dose of exosomes overexpressing CD24 (Experimental): The patients will receive the dose of 10^10 exosomes overexpressing CD24
  Interventions: Drug: CovenD24

INTERVENTIONS:
Drug: CovenD24 — The drug will be administrated once daily for 5 days
  Other Names: Exo-CD24

SUMMARY:
This is a phase II randomized, single-blind dose study to evaluate the safety and efficacy of exosomes overexpressing CD24 of two doses, Dose 1 - 10^9 exosome particles (per dose) versus Dose 2 - 10^10 exosome particles (per dose), to prevent clinical deterioration in patients with Moderate or Severe COVID-19 infection.

DETAILED DESCRIPTION:
The study population will include patients with moderate or severe COVID-19 and laboratory markers predictive of the cytokine storm, who have provided an informed consent.

90 patients will be randomized in a 1:1 ratio to receive either 109 exosome particles (45 patients) or 1010 exosome particles (45 patients).

The exosomes will be diluted in normal saline for inhalation via mouthpiece nebulization, administered once daily (QD) for 5 days.

Study treatments will be given as an add-on to the standard of care. Following the 5 days of treatment, patients will remain in follow-up for 23 additional days. In case of hospital discharge before the full follow-up planned, the patient will be required to return to the site for completion of all study assessments.

ELIGIBILITY:
Inclusion Criteria:

1. A COVID-19 diagnosis confirmed with a SARS-CoV-2 infection positive polymerase chain reaction (PCR) within 30 days of screening.
2. Age 18-80 years.
3. Severity of disease according to the following criteria (at least one clinical parameter and one laboratory parameter are required):

   a. Clinical and Imaging-based evaluation i. Respiratory rate > 23/min and < 30/min ii. SpO2 at room air ≤94% and ≥90% iii. Bilateral pulmonary infiltrates >25% within 24-48 hours or a severe deterioration compared to imaging at admission.

   b. Evidence of an exacerbated inflammatory process i. LDH > 300 U/L or what is the upper limit for normal per age ii. CRP >25 mg/L iii. Ferritin >500 ng/ml iv. Lymphocytes <800 cells/mm3 v. D-dimers > 500ng/ml
4. Willing and able to sign an informed consent.

Exclusion Criteria:

1. Any concomitant illness that, based on the judgment of the Investigator might affect the interpretation or the results of the study (i.e., immunodeficiency).
2. Mechanically-ventilated patient or patient who will probably require ICU admission or mechanical ventilation within 24 hours from enrolment, according to the Investigator's judgment.
3. Previous complete or partial vaccination for SARS-CoV-2.
4. Pregnancy [positive urine pregnancy test (women of childbearing potential only)] or breastfeeding.
5. Participation in any other Interventional study in the last 30 days
6. Active cancer.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-06-09 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Collection of serious adverse events | Through study completion, an average of 4 months
  * Incidence of treatment (dose)-related serious adverse events.
  * Incidence of all adverse events related or unrelated to the study treatment.
Proportion of patients related with Respiratory rate and SpO2 saturation | Through study completion, an average of 4 months
  * Proportion of patients with respiratory rate < 23/min for at least 24 hours, on Day 7.
  * Proportion of patients with SpO2 saturation >94%, on room air for at least 24 hours, on Day 7.
  * Proportion of patients with a decrease by 50% in either CRP/LDH/Fibrinogen/Ferritin/D-dimers from baseline to Day 7.

SECONDARY OUTCOMES:
Improvement of COVID19 status from severe to moderate | Through study completion, an average of 4 months
  • Rate of categorical and absolute score improvement of COVID-19 status on Day 7 improving from "Severe" to at least "Moderate" or from "Moderate" to "Moderate-Mild"
Time to recovery | Through study completion, an average of 4 months
  • Time to recovery, measured from enrolment (Day 1) to recovery or last follow-up (Day 28).
Death rate | Through study completion, an average of 4 months
  • Death rate at end of study (Day 28)
No need for mechanical ventilation | Through study completion, an average of 4 months
  • Proportion of patients with no mechanical ventilation (ECMO, NIV, high flow) on Day 7.
Patients status regarding haemodynamic instability | Through study completion, an average of 4 months
  • Proportion of patients with haemodynamic instability or requiring vasopressors on Day 7.
Oxygen saturation | Through study completion, an average of 4 months
  • Change in the SpO2/FiO2 ratio on Day 7.
Time to death or respiratory failure | Through study completion, an average of 4 months
  • Time to death or respiratory failure (defined as an arterial oxygen pressure (PaO2) of <60 mmHg and/or an arterial carbon dioxide pressure (PaCO2) of >45 mmHg, or the need for mechanical ventilation, ECMO, non-invasive ventilation, or high-flow oxygen devices) within 28 days of the study period (Day 1 to Day 28).
Hospital discharge time | Through study completion, an average of 4 months
  • Hospital discharge time within 28 days of the study period, calculated from the day of randomization (Day 1) to discharge or last follow-up (Day 28), whichever comes first.
No of patients that will need Intensive Care Unit | Through study completion, an average of 4 months
  • Proportion of patients requiring admission to an Intensive-Care Unit (ICU) on Day 7.
No of patients with respiratory rate < 23/min | Through study completion, an average of 4 months
  • Proportion of patients with respiratory rate < 23/min for 24 hours at every visit until Day 28, inclusive.
No of patients with change in respiratory change | Through study completion, an average of 4 months
  • Proportion of patients with change [decrease/no change (±2 breaths/min)/improvement] in respiratory rate from baseline to Day 7.
No of patients with SpO2 >94% | Through study completion, an average of 4 months
  • Proportion of patients with SpO2 >94% on room air, for at least 24 hours at every visit until Day 28, inclusive.
No of patients with change in oxygen saturation | Through study completion, an average of 4 months
  • Proportion of patients with change [decrease/no change (±2 %)/improvement] in SpO2 saturation from baseline to Day 7.
No of patients with change in lymphocyte count | Through study completion, an average of 4 months
  • Proportion of patients with an increase of 25% in the absolute lymphocyte count, sustained for ≥24 hours on Day 7.
Changes in absolute lymphocyte count | Through study completion, an average of 4 months
  • Change in absolute lymphocyte count from baseline to Day 7.
No of patients with changes in the neutrophil-to-lymphocyte ratio | Through study completion, an average of 4 months
  • Proportion of patients with a decrease of 20% in the neutrophil-to-lymphocyte ratio (NLR), sustained for ≥24 hours on Day 7.
Changes in the neutrophil-to-lymphocyte ratio | Through study completion, an average of 4 months
  • Change in NLR from baseline to Day 7.
No of patients with changes in disease severity | Through study completion, an average of 4 months
  • Percentage of patients within each severity rating on the ordinal scale within 28 days of the study period (Day 1 to Day 28).
Time of disease improvement | Through study completion, an average of 4 months
  • Time to improvement in the categorical and ordinal scale, measured from randomization (Day 1) to last study follow-up (Day 28).
Changes in COVID-19 clinical severity | Through study completion, an average of 4 months
  • Change in the COVID-19 clinical severity from baseline [before-treatment assessment (Screening/Day 1)] up to Day 28.
Changes in common COVID-19 related symptoms | Through study completion, an average of 4 months
  • Change from baseline of 14 Common COVID-19-Related Symptoms, as assessed through an Investigator interview.
Changes in supplemental oxygen over time | Through study completion, an average of 4 months
  • Change in the flow rate of supplemental oxygen administration over time.
Duration of oxygen administration | Through study completion, an average of 4 months
  • The duration of supplemental (non-invasive) oxygen administration.

CONTACTS AND LOCATIONS:
Overall Officials: Sotirios Tsiodras, Prof, Principal Investigator — Attikon University Hospital, Athens, Greece
Locations (3):
- Greece (3):
  - 3rd Department of Medicine, "Sotiria" Thoracic Diseases General Hospital of Athens, Athens, Attica
  - 7th Respiratory Medicine Department, "Sotiria" Thoracic Diseases General Hospital of Athens, Athens, Attica
  - Attikon University Hospital, Athens, Attica

IPD SHARING:
Plan to Share IPD: No